CLINICAL TRIAL: NCT06548880
Title: Investigation of the Effectiveness of Online Exercise Training in Geriatric Population Whose Daily Life Activity Level Decreased During COVID-19 Pandemic
Brief Title: Effectiveness of Online Exercise Training in Geriatric Population During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Collaborators: Istanbul Gedik University (Other)
Responsible Party: Principal Investigator, Sıla YILMAZ, Lecturer, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-714577430500104202121124-255
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-08

CONDITIONS: Aging; Falling; Dependence; Inactivity, Physical
Keywords: COVID-19; activities of daily living; geriatrics; telerehabilitation
MeSH Terms: conditions — Sedentary Behavior; COVID-19

STUDY DESIGN:
Intervention Model Description: 10 participants were included in the study group, and 10 participants were included in the control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Participants in the study group have received an online exercise training with a structured exercise program including range of motion, stretching, and, to train full body, low intensity aerobic exercises, once a week for 10 weeks, each lasting 60 minutes.
  Interventions: Other: Structured exercise program
- Control group (No Intervention): Participants in the control group were asked to maintain their daily physical activity routine.

INTERVENTIONS:
Other: Structured exercise program — The intervention applied in this research has an online exercise training conducting with a structured exercise program including different types of exercise which are range of motion, stretching and low intensity aerobic exercises. The exercise program continued with sessions each lasting 60 minutes, once a week for 10 weeks.
  Arms: Study group

SUMMARY:
The aim of this study is to investigate the effectiveness of online exercise training in geriatric population whose daily life activity level decreased during COVID-19 pandemic.

The main questions it aims to answer are:

* Does online exercise training improve quality of life in the geriatric population whose daily life activity levels have decreased during the COVID-19 pandemic?
* Does online exercise training improve sleep quality in the geriatric population whose daily life activity levels have decreased during the COVID-19 pandemic?
* Does online exercise training affect depression status in the geriatric population whose daily life activity levels have decreased during the COVID-19 pandemic?
* Does online exercise training reduce the risk of falls by improving balance and functional independence in geriatric population whose daily life activity levels have decreased during the COVID-19 pandemic?
* Does online exercise training improve posture in geriatric population whose daily life activity levels have decreased during the COVID-19 pandemic?

Research data were collected by Sociodemographic Information Form, 36-Item Short Form Survey, The Pittsburgh Sleep Quality Index, Geriatric Depression Scale, Timed Up & Go Test, and New York Posture Rating Chart.

While no application was given to the control group, study group has received an online exercise training with a structured exercise program including range of motion, stretching, and, to train full body, low intensity aerobic exercises, once a week for 10 weeks, each lasting 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being over 65 years old

Exclusion Criteria:

* Having mental retardation at a level that prevents communication
* Having an uncontrollable heart and hypertension problem
* Being receiving medical treatment or rehabilitation for balance that may affect the balance level
* Having osteoporosis at a level where exercise can be considered risky
* Having a health problem where exercise is considered contraindicated

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
balance | This outcome was evaluated twice, before starting the exercise program and after completing the exercise program.
  To determine fall risk and measure the progress of balance, sit to stand and walking, Timed-Up and Go Test was used. This is a simple screening test that is a sensitive and specific measure of probability for falls among older adults. An older adult who takes ≥12 seconds to complete the test is at risk for falling. The results of the Timed-Up and Go Test were obtained in seconds. This primary outcome was evaluated by interpreting these results.
mobility | This outcome was evaluated twice, before starting the exercise program and after completing the exercise program.
  To determine fall risk and measure the progress of balance, sit to stand and walking, Timed-Up and Go Test was used. This is a simple screening test that is a sensitive and specific measure of probability for falls among older adults. An older adult who takes ≥12 seconds to complete the test is at risk for falling. The results of the Timed-Up and Go Test were obtained in seconds. This primary outcome was evaluated by interpreting these results.

SECONDARY OUTCOMES:
sleep quality | This outcome was evaluated twice, before starting the exercise program and after completing the exercise program.
  This outcome was evaluated by The Pittsburgh Sleep Quality Index. This is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score. Each item is weighted on a 0-3 interval scale. The global score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
depression status | This outcome was evaluated twice, before starting the exercise program and after completing the exercise program.
  This outcome was evaluated by Geriatric Depression Scale. According to the results of this questionnaire, a higher score is considered an indicator of more severe depression.
posture | This outcome was evaluated twice, before starting the exercise program and after completing the exercise program.
  This outcome was evaluated by New York Posture Rating Chart. This test includes a set of three figure drawings for each of different body alignment segments contributing to overall postural alignment. According to the results of this test, a higher score is considered an indicator of good posture.
QoL | This outcome was evaluated twice, before starting the exercise program and after completing the exercise program.
  This outcome was evaluated by 36-Item Short Form Survey. This questionnaire evaluates 8 basic concepts related to health with 36 questions. Item scores for each quality of life area are coded and placed on a scale of 0-100 (0 is the worst, 100 is the best) using algorithms.

CONTACTS AND LOCATIONS:
Overall Officials: Gönül ERTUNÇ GÜLÇELİK, Ph.D., Study Chair — Kocaeli University; Sıla YILMAZ, M.Sc., Study Director — Medipol University; Fatma Nur DÜLGER, Miss, Principal Investigator — Medipol University; Elvan EKİNCİ, Miss, Principal Investigator — İstanbul Gedik University
Locations (1):
- Medipol University, Istanbul, Turkey (Türkiye)